CLINICAL TRIAL: NCT03819751
Title: MRI-targeted Biopsy of the Prostate: a Prospective Comparison of Software-based Fusion Versus Visual (Cognitive) Registration in the Accuracy of Clinically Significant Prostate Cancer Detection
Brief Title: MRI-targeted Biopsy of the Prostate: Software Versus Visual Registration in the Accuracy of Prostate Cancer Detection
Acronym: PROSOVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s.nr
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Prostate Neoplasm
Keywords: prostatic neoplasms; biopsy; Multimodal Imaging; prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients receive both types of biopsy. Patients are randomized with one half having visual registration first and the other half having software registration first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI-targeted prostate biopsy (Other): Participants receive both type of MRI-targeted biopsy. Patients are randomized with one half having visual registration first and the other half having software registration first.
  Interventions: Procedure: MRI-targeted prostate biopsy

INTERVENTIONS:
Procedure: MRI-targeted prostate biopsy — All participants receive traditional cognitive/visual registration biopsy and the above mentioned MRI/TRUS fusion biopsy (also known as software registration biopsy)
  Other Names: MRI/TRUS fusion biopsy with Philips Percunav

SUMMARY:
With the general acceptance of MRI and technical advances in biopsy technique of the prostate, new questions arise concerning the selection of patients, the approach, the appropriate technique, the lesions to target and the number of biopsies. The purpose of this study is to address these issues in men suspicious of having prostate cancer and without prior biopsies.

DETAILED DESCRIPTION:
Trial Design: This is a prospective, single center, comparative, diagnostic study of two biopsy techniques. All men aged 50 to 75 years with clinical suspicion of PCa (elevated prostate specific antigen (PSA) levels in blood and/or abnormal digital rectal examination) and an MRI with suspicious lesion(s) (presence of PI-RADS 3-5 lesion) will be included. Participants receive both types of biopsy, but will be randomized concerning the order of the biopsy. All men will also receive traditional systematic biopsies. Treatment and further follow-up is according to EAU guidelines. Data of treatment and follow-up will be retrieved till 2 years after initial MRI-visit.

Sample Size: Based on McNemar test for the comparison between the accuracy of the two biopsy techniques, the required sample size is estimated on 96 patients.

Assessment of efficacy: Efficacy of software and visual registration biopsy will be determined by histopathology: cancer core length (actual length and percentage) and comparison with systematic biopsy as reference standard.

Direct access to source data and documents: The investigator(s) and the institution(s) will permit trial-related monitoring, audits, EC review, and regulatory inspections (where appropriate) by providing direct access to source data and other documents (i.e. patients' case sheets, blood test reports, X-ray reports, histology reports, etc.).

Data handling and management: All data collected during the study remain confidential and according to the GDPR regulation. Data of the participants will be retrieved from their electronic patient files. Each participant will be given a unique identification number. When data are coded, there continues to be a link between the data and the individual who provided it. The research team is obligated to protect the data from disclosure outside the research according to the terms of the research protocol and the informed consent document. The subject's name or other identifiers should be stored separately (site file) from their research data and replaced with a unique code to create a new identity for the subject. Note that coded data are not anonymous. All data is collected and stored electronically by the principal investigator and co-investigators.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study by giving written informed consent.
* male subjects aged between 50 to 75 years.
* with a clinical suspicion of PCa: elevated prostate specific antigen (PSA) levels in blood and/or abnormal digital rectal examination (DRE).
* good health condition based on medical history, physical examination and vital sign measurements.
* with target lesion on dedicated MRI of the prostate (PI-RADS 3 to 5).

Exclusion Criteria:

* has a prior history of prostate cancer.
* had prior prostate biopsy.
* has a contra-indication for MRI (claustrophobia, non-compatible metallic implants).
* has evidence of lymph nodes involvement on prostate MRI or abdominal CT
* has evidence of bone metastasis on bone scan.
* has a prior history of hip prosthesis, pelvic radiation therapy or androgen deprivation therapy
* unable to perform transrectal ultrasound due to prior rectal surgery or active rectal diseases (rectitis, …)
* has any condition, physical, mental, familial or sociological, that could impede compliance with the study protocol and further follow-up. This is not an absolute contra-indication, but should be discussed with patient prior to registration in the trial.

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants need to have a prostate.
Enrollment: 96 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the two MR-guided registration techniques (visual and software-based) in the detection of clinically significant prostate cancer | From MRI-visit till results of radical prostatectomy is known or till up to 2 years after MRI-visit
  Assessment of the detection rate of clinically significant prostate cancer of software registration biopsy and visual registration biopsy, using traditional TRUS-guided systematic biopsy, whole mount radical prostatectomy specimen and follow-up as reference.

SECONDARY OUTCOMES:
Analysis of the performance of software versus visual registration biopsy in subgroups | From MRI-visit till results of radical prostatectomy is known or till up to 2 years after MRI-visit
  Assessment of the performance of software registration biopsy and visual registration biopsy in the detection of clinically significant cancer in :
  * lesions in small volume prostates (<50 gram) versus large volume prostates (>50 gram).
  * transitional zone versus peripheral zone lesions
  * basal versus apical lesions
  * small (max. diameter < or = 10 mm) versus large lesions (max. diameter > 10 mm)
  * intermediate suspicious lesions (PI-RADS 3) versus highly suspicious lesions (PI-RADS 4-5).
Added value of systematic biopsies | From MRI-visit till results of radical prostatectomy is known or till up to 2 years after MRI-visit
  Assessment of the added value of systematic biopsies on top of MRI-targeted biopsy of PI-RADS 3, 4 and 5 lesions. Compare MRI-targeted + systematic biopsies versus MRI-targeted biopsies alone in T-staging and therapy options.
Discriminative features of PI-RADS 3 lesions on MRI | From MRI-visit till results of radical prostatectomy is known or till up to 2 years after MRI-visit
  Lesion diameters, shape, intensity on T2 and aspect, ADC-values on ADC-map will be measured to identify possible discriminative features of 'malignant' s "benigne" PI-RADS 3 lesions.
Features of prostate cancer differentiation grade on MRI | From MRI-visit till results of radical prostatectomy is known or till up to 2 years after MRI-visit
  Measure ADC-value to differentiate prostate cancer differentiation grade.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Mai, MD, Principal Investigator — University Hospital Leuven, Department of Radiology
Locations (1):
- UZ Leuven, Leuven, Vlaams-brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Futterer JJ, Briganti A, De Visschere P, Emberton M, Giannarini G, Kirkham A, Taneja SS, Thoeny H, Villeirs G, Villers A. Can Clinically Significant Prostate Cancer Be Detected with Multiparametric Magnetic Resonance Imaging? A Systematic Review of the Literature. Eur Urol. 2015 Dec;68(6):1045-53. doi: 10.1016/j.eururo.2015.01.013. Epub 2015 Feb 2. PMID 25656808
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Kasivisvanathan V, Emberton M, Moore CM. MRI-Targeted Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 Aug 9;379(6):589-590. doi: 10.1056/NEJMc1807507. No abstract available. PMID 30089067
- [Background] Moore CM, Robertson NL, Arsanious N, Middleton T, Villers A, Klotz L, Taneja SS, Emberton M. Image-guided prostate biopsy using magnetic resonance imaging-derived targets: a systematic review. Eur Urol. 2013 Jan;63(1):125-40. doi: 10.1016/j.eururo.2012.06.004. Epub 2012 Jun 13. PMID 22743165
- [Background] Logan JK, Rais-Bahrami S, Turkbey B, Gomella A, Amalou H, Choyke PL, Wood BJ, Pinto PA. Current status of magnetic resonance imaging (MRI) and ultrasonography fusion software platforms for guidance of prostate biopsies. BJU Int. 2014 Nov;114(5):641-52. doi: 10.1111/bju.12593. Epub 2014 May 22. PMID 24298917
- [Background] Wysock JS, Rosenkrantz AB, Huang WC, Stifelman MD, Lepor H, Deng FM, Melamed J, Taneja SS. A prospective, blinded comparison of magnetic resonance (MR) imaging-ultrasound fusion and visual estimation in the performance of MR-targeted prostate biopsy: the PROFUS trial. Eur Urol. 2014 Aug;66(2):343-51. doi: 10.1016/j.eururo.2013.10.048. Epub 2013 Nov 8. PMID 24262102
- [Background] Puech P, Rouviere O, Renard-Penna R, Villers A, Devos P, Colombel M, Bitker MO, Leroy X, Mege-Lechevallier F, Comperat E, Ouzzane A, Lemaitre L. Prostate cancer diagnosis: multiparametric MR-targeted biopsy with cognitive and transrectal US-MR fusion guidance versus systematic biopsy--prospective multicenter study. Radiology. 2013 Aug;268(2):461-9. doi: 10.1148/radiol.13121501. Epub 2013 Apr 11. PMID 23579051
- [Background] Moore CM, Kasivisvanathan V, Eggener S, Emberton M, Futterer JJ, Gill IS, Grubb Iii RL, Hadaschik B, Klotz L, Margolis DJ, Marks LS, Melamed J, Oto A, Palmer SL, Pinto P, Puech P, Punwani S, Rosenkrantz AB, Schoots IG, Simon R, Taneja SS, Turkbey B, Ukimura O, van der Meulen J, Villers A, Watanabe Y; START Consortium. Standards of reporting for MRI-targeted biopsy studies (START) of the prostate: recommendations from an International Working Group. Eur Urol. 2013 Oct;64(4):544-52. doi: 10.1016/j.eururo.2013.03.030. Epub 2013 Mar 20. PMID 23537686